CLINICAL TRIAL: NCT00083291
Title: Pilot Study of Helicobacter Pylori and Ocular Surface Disease
Brief Title: Helicobacter Pylori and Dry Eye
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040190; 04-EI-0190
Record Dates: First submitted 2004-05-18; First posted 2004-05-18 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-03

CONDITIONS: Helicobacter Infections
Keywords: Dry Eyes; Conjunctiva; Infection; Antibodies; Inflammation; Ocular Surface Disease; Helicobacter Pylori
MeSH Terms: conditions — Helicobacter Infections; Dry Eye Syndromes; Infections; Inflammation

SUMMARY:
This study will examine whether infection with Helicobacter pylori bacteria may cause inflammation of the eye's surface. Although most people who are infected with H. pylori do not have symptoms, the bacteria can cause several diseases, including gastritis-stomach inflammation, stomach ulcers or, rarely, stomach cancer, and certain types of lymphoma. H. pylori has also been associated with autoimmune disorders, in which the patient's immune system attacks the body's own tissues.

People who have been infected with H. pylori, with and without dry eye, may be eligible for this study. Candidates are screened with a medical history, a blood test to determine H. pylori infection, and an eye examination. The examination includes measurements of visual acuity, eye pressure, and tear production. To measure the amount of tear production, a small piece of filter paper is inserted over the eyelid on the side and collects tears over a 5-minute period. Drops of two colored dyes (orange and green) are placed in the eyes to see if there are any dry areas. Screening also includes examination of the pupils and eye movements, the lens, and the back of the eye, including the retina.

Participants will also have a few cells collected from the surface of the eye. After the eyes are numbed with anesthetic eye drops, a swab (like a Q-tip) is rolled over the surface of the white part of the eye to collect small samples of the superficial layer of the conjunctiva - a transparent membrane covering the eyeball. The specimens are analyzed by special laboratory techniques to determine whether H. pylori has infected the eye.

DETAILED DESCRIPTION:
Helicobacter pylori, one of the world's most prevalent pathogens, is a spiral-shaped, catalase-positive, Gram-negative rod with 4-6 sheathed flagella attached to one pole which allow for motility. The prevalence of H. pylori infection in humans is high; 50% of those over the age of 60 are infected. H. pylori infection causes chronic gastric inflammation, ulcer disease and gastric carcinoma. Further, chronic antigenic stimulation driven by H. pylori infection has been linked to the development of gastric mucosa associated lymphoid tissue (MALT) lymphoma. Infection with H. pylori induces a vigorous immune response resulting in the presence of local and systemic antibodies. H. pylori-specific immunoglobulin G antibodies present in serum, plasma, whole blood, saliva, gastric juice and urine have each been used to successfully detect the presence of infection in adults. The sensitivity and specificity of serological tests range from 80% to 95% depending upon the assay used. H. Pylori infection is characteristically associated with a vigorous inflammatory response and we have recently identified H. Pylori DNA in conjunctival MALT lymphoma using molecular diagnostic techniques. Ocular surface inflammation is a cardinal feature of keratoconjunctivitis sicca. Since we identified H. Pylori DNA in conjunctival MALT lymphoma we hypothesize that chronic infection may also be capable of triggering chronic ocular surface inflammation as seen in keratoconjunctivitis sicca. The purpose of this pilot study is to determine whether H. pylori DNA is detectable in the conjunctiva of seropositive KCS patients.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients with ocular surface disease including aqueous or evaporative tear deficiency who are seropositive for H. pylori will be eligible. Controls will be adults without ocular surface disease who are seropositve for H. pylori.

EXCLUSION CRITERIA:

None listed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 2004-05; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Patel P, Mendall MA, Carrington D, Strachan DP, Leatham E, Molineaux N, Levy J, Blakeston C, Seymour CA, Camm AJ, et al. Association of Helicobacter pylori and Chlamydia pneumoniae infections with coronary heart disease and cardiovascular risk factors. BMJ. 1995 Sep 16;311(7007):711-4. doi: 10.1136/bmj.311.7007.711. PMID 7549683
- [Background] Weger M, Haas A, Stanger O, El-Shabrawi Y, Temmel W, Maier R, Berghold A, Haller-Schober EM. Chlamydia pneumoniae seropositivity and the risk of nonarteritic ischemic optic neuropathy. Ophthalmology. 2002 Apr;109(4):749-52. doi: 10.1016/s0161-6420(01)01031-4. PMID 11927434
- [Background] Kalayoglu MV, Galvan C, Mahdi OS, Byrne GI, Mansour S. Serological association between Chlamydia pneumoniae infection and age-related macular degeneration. Arch Ophthalmol. 2003 Apr;121(4):478-82. doi: 10.1001/archopht.121.4.478. PMID 12695244